CLINICAL TRIAL: NCT03928249
Title: Therapeutic Intervention of Eriocitrin in Reducing Hyperglycemia in Pre-diabetic Subjects: Double-blind, Randomized, Placebo-controlled Crossover Clinical Trial
Brief Title: Therapeutic Intervention of Eriocitrin in the Reduction of Hyperglycemia in Pre-diabetic Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: São Paulo State University (Other)
Responsible Party: Principal Investigator, Thais Cesar, Principal Investigator, São Paulo State University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: SaoPSU12
Record Dates: First submitted 2019-04-17; First posted 2019-04-26 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Pre Diabetes
Keywords: Eriocitrin; Citrus bioflavonoids; Flavanone; Pre-diabetes; Blood glucose
MeSH Terms: conditions — Glucose Intolerance | interventions — eriocitrin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Grupo A (Active Comparator): Group A (n = 20) will receive 200 mg / d of eriocitrin for 12 weeks, washout for 2 weeks and then receive 200 mg / d of placebo for 12 weeks
  Interventions: Dietary Supplement: Eriocitrin
- GRUPO B (Placebo Comparator): group B (n = 20) will receive 200 mg / d placebo for 12 weeks with washout for 2 weeks and then receive 200 mg / d placebo for 12 weeks
  Interventions: Dietary Supplement: Eriocitrin

INTERVENTIONS:
Dietary Supplement: Eriocitrin — A crossover, double-blind, randomized, placebo-controlled clinical study with a duration of 26 weeks will be performed. All individuals and the principal investigator will remain blind to treatment until all analyzes are completed.
  Participants will be invited to attend 12-hour fasting to measure glucose levels, glycated hemoglobin and to perform the glucose tolerance test, in addition to an individual interview (Appendix B) to confirm eligibility according to the inclusion and exclusion criteria . The collection of blood and the glycemic curves will be performed at the beginning of the first, 12th, 14th and 26th week in the Laboratory of Clinical Analyzes ( Araraquara)
  At the beginning of the first, 12th, 14th and 26th week the following anthropometric parameters will be evaluated: body weight (kg), muscle mass (kg), fat mass (kg), body fat (%) (InBody 720, Biospace, Tokyo, Japan ) and waist-hip ratio.

SUMMARY:
Supplementation with citrus bioflavonoids (hesperidin, naringin, diosmin and eriocitrin, among others) has been associated with an improvement in the glycidic and lipid profile, reduction of insulin resistance and systemic inflammation, and reduction of endothelial damage. This study aims to evaluate the effects of eriocitrin supplementation on the metabolic parameters of pre-diabetic individuals. Participants will be adults with pre-diabetes who will receive 200 mg / d of eriocitrin. Before, during and after treatment, anthropometric measures (weight, body composition and circumferences), biochemical (lipid and glucose profile, inflammatory parameters, endothelial markers, liver function, renal function) will be evaluated. Metabolic parameters that constitute risk factors for diabetes and associated chronic diseases are expected to be improved by supplementation with eriocitrin.

DETAILED DESCRIPTION:
Individuals aged 35-60 years and who present at least one of the following criteria: (1) increased fasting blood glucose from 6.1 to 7.0 mmol / L, (2) decreased glucose tolerance of 7 , 8 to 11.1 mmol / L, and (3) glycated hemoglobin with values between 5.7 and 6.4% 10 will be eligible to participate in this study. The exclusion criteria will be to use hypoglycemic, hypolipidemic drugs, dietary supplements (vitamins, minerals, bioflavonoids, prebiotics, probiotics or other bioactive compounds), exercise intensely (more than 10 hours per week), history of cardiovascular diseases , diabetes mellitus, liver and kidney disease.

The selected individuals will be distributed randomly in 2 groups through random number generator program. Group A (n = 20) will receive 200 mg / d of eriocitrin for 12 weeks, with washout for 2 weeks and then receive 200 mg / d of placebo for 12 weeks; group B (n = 20) will receive 200 mg / d placebo for 12 weeks with washout for 2 weeks and then receive 200 mg / d placebo for 12 weeks.

The primary endpoint will be fasting blood glucose, blood glucose 2 hours after oral glucose tolerance test (GTTO), and HbA1c. The secondary endpoint will be insulin, HOMA-IR, total cholesterol, triglycerides, HDL-cholesterol, LDL-cholesterol, ALP, yGT, AST, ALT, TNF-α, IL-6, CRP, body weight, body mass index BMI), muscle mass, fat mass, body fat and waist-hip ratio, and macronutrient intake.

ELIGIBILITY:
Inclusion Criteria:

* 35-60 years
* Increased fasting blood glucose from 6.1 to 7.0 mmol / L or,
* Decreased glucose tolerance of 7 , 8 to 11.1 mmol / L or,
* Glycated hemoglobin with values between 5.7 and 6.4%

Exclusion Criteria:

* Use hypoglycemic, hypolipidemic drugs,
* Use dietary supplements (vitamins, minerals, bioflavonoids, prebiotics, probiotics or other bioactive compounds),
* Exercise intensely (more than 10 hours per week)
* History of cardiovascular diseases , diabetes mellitus, liver and kidney disease.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-10-22 (Actual)

PRIMARY OUTCOMES:
Fasting glycemia | 0-12-18-26 week
  Changes in serum glycemia concentration before and after administration of the intervention/placebo

SECONDARY OUTCOMES:
Rate of change in plasma glucose concentration | 0-12-18-26 week
  Changes in serum 2 hours after oral glucose tolerance test (mg/dL) before and after administration of the intervention / placebo
Rate of change in plasma HbA1c | 0-12-18-26 week
  Changes in serum HbA1c (%) before and after administration of the intervention / placebo
Rate of change in plasma insulin concentration | 0-12-18-26 week
  Changes in serum insulin (µU/mL) before and after administration of the intervention / placebo
Rate of change in plasma lipid concentration | 0-12-18-26 week
  Changes in serum cholesterol (mg/dL), triglycerides (mg/dL),HDL-C(mg/dL), LDL-C(mg/dL) before and after administration of the intervention/placebo
Rate of change in plasma hepatic enzymes | 0-12-18-26 week
  Changes in ALT (U/L), AST (U/L), ALP (U/L), GGT (U/L) before and after administration of the intervention / placebo
Rate of change in plasma inflammatory parameters | 0-12-18-26 week
  Changes in CRP (mg/dL), TNF-a (mg/dL), IL-6 (mg/dL) before and after administration of the intervention / placebo
Rate of change in anthropometric parameters | 0-12-18-26 week
  Changes in body weight (Kg), muscle mass (Kg), fat mass (Kg) before and after administration of the intervention / placebo

CONTACTS AND LOCATIONS:
Overall Officials: Thais B Cesar, Phd, Principal Investigator — Sao Paulo State University "Julio de Mesquita Filho"
Locations (1):
- Sao Paulo State University "Julio de Mesquita Filho", Araraquara, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No